CLINICAL TRIAL: NCT03862560
Title: Evaluación Del Rendimiento físico y asimetrías Funcionales en el fútbol Femenino
Brief Title: Evaluation of Physical Performance and Functional Asymmetries in Female Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, José A. Casajús, Senior Lecturer, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C.P. - C.I. PI19/039
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Resistance Training; Inter-limb Asymmetries; Athletic Performance
Keywords: Soccer; Female; Lower limb asymmetries; Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Female soccers that perform a strength training
  Interventions: Other: Strength training program
- Control group (No Intervention): Female soccers that do not perform a strength training

INTERVENTIONS:
Other: Strength training program — Strength training program in female soccer players
  Arms: Experimental group

SUMMARY:
Worldwide, soccer has grown increasingly popular among female players. According to the Women´s Football Survey of the Fédération Internationale de Football Association (FIFA), there were more than 30 million registered women soccer players in 2014. Elite female soccer players cover approximately a total distance of 10 km with 1.7 km completed at high-speed (>18 km/h-1), between 1350 and 1650 changes of activity like passing, dribbling, tackling and trapping and 5.1 and 31.2 repeated sprinting and high intensity bouts, respectively. Thus, it seems that those strategies addressed to improve such high-intensity activities should be considered a priority for female soccer players.

Different training methods to improve soccer specific variables have been developed such as, high-intensity interval training, resisted sprint training, strength training or plyometric training. Whilst individual training interventions have been shown to produce enhancements in measures of athletic performance for soccer players, there is a paucity of studies looking at the effectiveness of strength and power training specifically on performance measures in female soccer populations.

Unilateral strength asymmetry can be a risk factor of musculoskeletal injuries. In recent years, inter-limb asymmetries have been included in battery tests performed by different soccer clubs due to their relation with lower-limb injuries. Few studies have analysed the change of an intervention on inter-limb asymmetry in female soccer players, hence, more studies for this population are warranted.

The main aim of this research project is therefore, to evaluate the effect of a physical intervention on the performance and inter-limb asymmetries of female soccer players.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, Healthy participant, from 12 to 20 years old, with a history of training at least 3 years.

Exclusion Criteria:

* Non-caucasian, injury.

Ages: 12 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Jumping in centimeters | Change from baseline in jumping height at 12 weeks
  Jumping height was assessed using a vertical countermovement jump, drop jump and standing broad jump with flight.
Velocity in seconds | Change from baseline in velocity at 12 weeks
  Running speed was evaluated by a 40-m sprint time (standing start) with 10-m, 20-m, 30-m split times.
Change of direction in seconds | Change from Baseline in change of direction at 12 weeks
  Change of direction ability was assessed by 180º change of direction and V-cut tests.
Inter-limb asymmetry in % | Change from Baseline in inter-limb asymmetry at 12 weeks
  Inter-limb asymmetry was calculated using the following formula : Inter-limb asymmetry = 100/Max Value (right and left)*Min Value (right and left)*-1+100.

CONTACTS AND LOCATIONS:
Locations (1):
- GENUD Research group (Growth, Exercise, NUtrition and Development), Zaragoza, Spain

REFERENCES:
- [Result] Hoff J, Helgerud J. Endurance and strength training for soccer players: physiological considerations. Sports Med. 2004;34(3):165-80. doi: 10.2165/00007256-200434030-00003. PMID 14987126
- [Result] Olsen OE, Myklebust G, Engebretsen L, Holme I, Bahr R. Exercises to prevent lower limb injuries in youth sports: cluster randomised controlled trial. BMJ. 2005 Feb 26;330(7489):449. doi: 10.1136/bmj.38330.632801.8F. Epub 2005 Feb 7. PMID 15699058
- [Result] Brumitt J, Heiderscheit BC, Manske RC, Niemuth PE, Rauh MJ. Lower extremity functional tests and risk of injury in division iii collegiate athletes. Int J Sports Phys Ther. 2013 Jun;8(3):216-27. PMID 23772338
- [Result] Kiani A, Hellquist E, Ahlqvist K, Gedeborg R, Michaelsson K, Byberg L. Prevention of soccer-related knee injuries in teenaged girls. Arch Intern Med. 2010 Jan 11;170(1):43-9. doi: 10.1001/archinternmed.2009.289. PMID 20065198